CLINICAL TRIAL: NCT05267665
Title: Family Involvement in Treatment for PTSD (FIT-PTSD): A Brief, Feasible Method for Enhancing Outcomes, Retention, and Engagement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBP-005-21S
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic stress disorder; PTSD; Veteran; Family treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Family members are randomly assigned to one of the following two groups: Brief Family Intervention (BFI) where they receive a 2-session intervention designed to help them better understand and support the Veteran's individual trauma-focused treatment, or no BFI where they do not receive the BFI sessions.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors are blind to the condition of the family member/Veteran
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFI (Experimental): Family members in this arm receive the 2-session BFI intervention.
  Interventions: Behavioral: Brief Family Intervention (BFI)
- No BFI (No Intervention): Family members in this arm do not receive the BFI sessions

INTERVENTIONS:
Behavioral: Brief Family Intervention (BFI) — A 2-session psychoeducational and skills-based family intervention.
  Arms: BFI

SUMMARY:
Although effective treatments for PTSD exist, high rates of treatment dropout and sub-optimal response rates remain common. Incorporating family members in treatment represents one avenue for improving outcomes and providing Veteran-centered care, and surveys of Veterans in outpatient VA PTSD care indicate that 80% desire family involvement. The VA has invested many years and millions of dollars on the dissemination of Cognitive Processing Therapy (CPT) and Prolonged Exposure (PE) for PTSD. A family-based intervention that complements these two first-line treatments would capitalize on existing treatment infrastructure while also potentially boosting outcomes and retention.

Preliminary testing of the proposed Brief Family Intervention (BFI) resulted in 50% less dropout from CPT/PE among Veterans whose family members received the BFI. There was also a large impact on PTSD symptoms at 16 weeks (d = 1.12) in favor of the BFI group. The goal of this study is to test the effectiveness of the BFI among a fully-powered sample. One hundred Veteran-family member dyads (n = 200) will be recruited. Veterans will be beginning a course of usual-care CPT or PE at one of two VA sites. Family members will be randomized to receive or not receive the BFI, a two-session psychoeducational and skills-based protocol. PTSD symptom severity and treatment retention will be the primary outcomes. Assessments will be conducted by independent evaluators at baseline, 6-, 12-, 18-, and 26-weeks. Veterans whose family members receive the BFI are expected to have lower dropout and a greater rate of change in their PTSD symptoms compared to Veterans whose family members do not receive the BFI. If the BFI is found to increase the effectiveness of and retention in CPT/PE, it will be a highly appealing option for incorporating families into Veterans' PTSD care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for Veterans will include:

* a current DSM-5 diagnosis of PTSD
* Veteran status
* willing to have a family member involved in the study
* has recently begun or is currently initiating individual CPT or PE (completed no more than 3 sessions of the protocol at the time of the baseline assessment)

  * If taking psychotropic medication, the Veteran must be on a stable dose for at least 30 days.

Inclusion criteria for family members will include:

* age 18 or older, family member of the Veteran (significant other, parent, adult child, sibling, etc.)
* currently having frequent contact with the Veteran (three or more times per week)

Exclusion Criteria:

Exclusion criteria for Veterans will include:

* current engagement in couple/family treatment with the identified family member participant
* current severe substance use disorder (mild/moderate use disorders will not be excluded; any level of nicotine or caffeine use disorder accepted)
* current psychosis or unstable bipolar disorder diagnosis
* high suicidal risk
* significant cognitive impairment

Exclusion criteria for family members will include:

* same as listed for Veterans. Additionally
* family members will NOT be permitted to participate if they meet criteria for current PTSD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Week 26
  Severity of PTSD symptoms. Minimum score is 0 (best possible, no symptoms) and maximum score is 80 (worst possible, highest symptoms).
Adequate treatment dose | Week 26
  Categorical evaluation of whether the participant received 8 or more on-protocol sessions of CPT or PE during their 26-week study participation period. Possible scores are 0 (meaning <8 sessions received; this is considered a poor outcome) or 1 (meaning 8 or more sessions received; this is considered a good outcome).
Treatment dropout | Week 26
  Categorical evaluation of whether the participant dropped out of treatment early. Possible scores are 0 (meaning participant did not drop out of treatment early; this is considered a good outcome) or 1 (meaning participant did drop out of treatment early; this is considered a poor outcome).

SECONDARY OUTCOMES:
Homework compliance | Week 26
  Compliance with assigned homework during treatment. Minimum score is 0 (worst possible), maximum score is 150 (best possible).
Quality of Life Inventory (QOLI) | Week 26
  Quality of life. Minimum score is -6 (worst possible), maximum score is 6 (best possible).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Thompson-Hollands, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (3):
- United States (3):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
An anonymous dataset that meets VA standards for disclosure to the public will be made available within 1 year of publication. Prior to distributions, a privacy officer at the primary site will certify that all datasets contain no PHI. The PI will create a de-identified dataset that will include all publication variables. To remove some PHI, loss of information may occur. The PI will replace any identifiable information with study-specific numbers. Data collected on age will be replaced by the PI with age categories to ensure data is in accordance with PHI requirements for people 85 years of age and older (if applicable).
Supporting Information: Study Protocol, ICF
Time Frame: An anonymous dataset that meets VA standards for disclosure to the public will be made available within 1 year of publication. The data will be made available until the data is destroyed according to the required timelines in the VA Record Control Schedule.
Access Criteria: Individual requesting access to the data will be required to complete an adequate Data Use Agreement.